CLINICAL TRIAL: NCT03719131
Title: A Randomized Phase 2 Study of Rituxan Hycela in Patients With Advanced Melanoma Undergoing Combination Immune Checkpoint Blockade With Nivolumab and Ipilimumab
Brief Title: Rituximab and Hyaluronidase Human in Patients With Advanced Melanoma Undergoing Nivolumab and Ipilimumab Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Kavita Dhodapkar, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00105605; NCI-2018-01804 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4457-18 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cutaneous Melanoma, Stage III; Cutaneous Melanoma, Stage IV; Stage III Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Rituximab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (standard of care) (Active Comparator): This is standard of care arm: induction with 4 cycles (21 days each) of Ipilimumab and nivolumab followed by continuation with nivolumab alone every month X1 year (13 doses).
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Arm B (rituximab, hyaluronidase human) (Experimental): This includes induction with 4 cycles of ipilimumab and nivolumab X 4 cycles followed by continuation with nivolumab alone every month for 1 year as in standard of care arm. Each induction cycle is 21 days and includes ipilimumab on day 1 plus nivolumab on day 1. In addition, patients will receive 4 weekly doses of Rituxan (first dose intravenously and then 3 weekly doses subcutaneously). First dose of Rituxan will be administered one week following the start of cycle 1 of ipilimumab and nivolumab. All treatments will have a +/-3 business day window for administration.
  Interventions: Drug: Nivolumab; Biological: Rituximab and Hyaluronidase Human; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Receive standard of care nivolumab therapy
  Other Names: Opdivo
Biological: Rituximab and Hyaluronidase Human — Given IV or SC
  Other Names: Rituxan Hycela
  Arms: Arm B (rituximab, hyaluronidase human)
Drug: Ipilimumab — Receive standard of care ipilimumab therapy
  Other Names: Yervoy

SUMMARY:
This phase II trial studies whether rituximab and hyaluronidase human (Rituxan Hycela) can prevent immune related adverse events in participants with stage III-IV melanoma that cannot be removed by surgery who are undergoing nivolumab and ipilimumab therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare rates for grade 3-4 immune-related adverse event (IRAE)s in the first 6 months in patients treated with combination checkpoint blockade (CCB) therapy (anti-CTLA4 and anti-PD1) as a part of standard of care for advanced melanoma who are treated with a single course of 4 weekly doses of rituximab and hyaluronidase human (Rituxan) therapy versus those who are not treated with Rituxan.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability (in terms of Rituxan-related adverse events) in patients with melanoma receiving CCB.

II. To compare objective response rate in patients receiving CCB therapy + Rituxan versus CCB therapy alone.

III. To compare 1 year overall and progression-free survival in patients receiving CCB therapy + Rituxan versus CCB therapy alone.

IV. To compare changes in cluster of differentiation 21lo (CD21lo) B cells in patients receiving CCB therapy + Rituxan versus CCB therapy alone.

V. To compare changes in T cells in patients receiving CCB therapy + Rituxan versus CCB therapy alone.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A: Participants receive standard of care ipilimumab and nivolumab therapy.

ARM B: Participants receive standard of care ipilimumab and nivolumab therapy. On day 2 of each cycle, participants also receive rituximab and hyaluronidase human intravenously (IV) or subcutaneously (SC) weekly starting week 1 for 4 doses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinically eligible to receive Food and Drug Administration (FDA) approved standard of care combination immune checkpoint therapy with ipilimumab and nivolumab for unresectable stage III or stage IV melanoma.
* No therapy with immune checkpoint inhibitors within 1 year prior to starting combination checkpoint therapy. Prior adjuvant ipilimumab, nivolumab, or pembrolizumab as single agent is allowed if greater than 1 year since last treatment and patient had no grade 3 or 4 toxicities from the checkpoint inhibitors. History of adjuvant interferon is allowed.
* Obtained within one week prior to randomization:

  * White blood count ≥ 3,000/µL
  * Absolute neutrophil count (ANC) ≥ 1,500/µL
  * Platelet count ≥ 100,000/µL
  * Hemoglobin ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN) or serum creatinine clearance (CrCl) ≥ 40 ml/min
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN (≤ 5 x ULN for patients with documented liver metastases)
  * Alkaline phosphatase ≤ 2 X ULN (≤ 5 X ULN for those with bone metastasis)
  * Total bilirubin ≤ 1.5 X ULN except those with direct bilirubin or Gilbert's syndrome
  * Serum lactate dehydrogenase (LDH) ≤ 10 X ULN

Exclusion Criteria:

* Allergy to rituximab, or any of the ingredients in rituximab injection or rituximab and hyaluronidase human injection.
* Patients with active central nervous system (CNS) metastatic disease or leptomeningeal disease. Patients with CNS metastatic disease that has been treated with surgical resection or stereotactic radiosurgery are eligible if lesions are stable for at least 4 weeks following therapy as determined by magnetic resonance imaging (MRI) scan done within one week of randomization.
* Prior therapy with immune checkpoint blocking antibodies (unless monotherapy given at least 1 year prior to starting combination therapy and no grade 3-4 toxicities while on monotherapy), vaccines or interleukin-2 (IL-2).
* Patients may have had prior systemic therapy in the adjuvant setting (e.g. interferon, proto-oncogene B-Raf [BRAF], or mitogen-activated protein-extracellular signal-regulated kinase [MEK] agents). Adjuvant ipilimumab, nivolumab, or pembrolizumab as single agent is allowed if greater than 1 year since last treatment and patient had no grade 3 or 4 toxicities from the checkpoint inhibitors.
* Women must not be pregnant or lactating. Must have negative urine or blood pregnancy test within 1 week of starting therapy.
* Patients with known human immunodeficiency virus (HIV) are ineligible.
* Patients with active Hepatitis B Virus (HBV) or Hepatitis C virus (HCV) are ineligible. -- ----Patients with prior history of, or serology suggestive of prior infection with Hepatitis B Virus (HBV) or Hepatitis C virus (HCV) are also ineligible.
* Patients with active, known or suspected autoimmune disorders including lupus and type I diabetes are ineligible. Patients with history of vitiligo, thyroiditis are eligible.
* Patients with active disease or history of inflammatory bowel disease are ineligible.
* Patients cannot be on corticosteroid therapy except as physiologic replacement therapy.
* Patients receiving ongoing corticosteroid therapy for autoimmune disorders are ineligible. Occasional steroid inhaler use or nasal spray are allowed. Patients receiving replacement doses of steroids for adrenal insufficiency are eligible.
* Patients must not have any serious underlying medical conditions or take medications that in the investigators opinion may interfere with compliance or interpretation of Immune-related adverse events (IRAEs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Dhodapkar, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Standard of Care) | Arm B (Rituximab, Hyaluronidase Human)
Started | 7 | 7
Completed | 6 | 5
Not Completed | 1 | 2
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Standard of Care) | Arm B (Rituximab, Hyaluronidase Human) | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Common Terminology Criteria (CTC) (Version [v]5.0) Grade 3 or Greater Immune-related Adverse Events
Description: All patients will be evaluable for toxicity from the time of their first treatment with ipilimumab/nivolumab. Investigators will review the toxicities, grade, and attribute each toxicity.
Time Frame: At 6 months after study start
Population: All patients were evaluated for toxicity from the time of their first treatment with ipilimumab/nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Standard of Care) | Arm B (Rituximab, Hyaluronidase Human)
Number analyzed (Participants) | 7 | 7
Participants | 4 | 1

2. Secondary Outcome: Rate of CTC (v5.0) Toxicity Related to Rituximab and Hyaluronidase Human
Description: as for outcome 1
Time Frame: Up to 4 weeks after study start
Reporting Status: Not Posted

3. Secondary Outcome: Objective Tumor Response
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune-related (ir)RECIST. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. Patients who exhibit objective disease progression prior to the end of cycle 1 will also be considered evaluable.
Time Frame: At 12 weeks and every 12 weeks thereafter up to 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Rate of Overall Survival
Description: Overall survival is defined as the duration of time from start of treatment to time of death or last follow-up, whichever occurs first.
Time Frame: From start of treatment up to 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Rate of Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death or last follow-up, whichever occurs first.
Time Frame: From start of treatment up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years and 4 months
Arm/Group | Arm A (Standard of Care) | Arm B (Rituximab, Hyaluronidase Human)
All-Cause Mortality (participants affected / at risk) | 1/7 | 2/7
Serious Adverse Events (participants affected / at risk) | 4/7 | 4/7
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Standard of Care) (N=7) | Arm B (Rituximab, Hyaluronidase Human) (N=7)
Hospitalization (Investigations) | 4 (8) | 4 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Standard of Care) (N=7) | Arm B (Rituximab, Hyaluronidase Human) (N=7)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Vestibular Disorder (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (4) | 1 (3)
Stabbing Lesion Pain (Back) (General disorders) | 1 (2) | 0 (0)
Rash/itching (arms and legs) (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Joint pain (General disorders) | 1 (2) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Fatigue (General disorders) | 4 (6) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (5) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 3 (7) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 2 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Hypoxia (Hospitalization) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
General Disorders and Administration Site Conditions (General disorders) | 1 (2) | 1 (6)
Nausea (Gastrointestinal disorders) | 3 (12) | 3 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (10)
Infusion related reaction (nivo reaction) (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fever (General disorders) | 4 (9) | 0 (0)
Cough (dry cough) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (General disorders) | 0 (0) | 1 (1)
AE Not Defined (Nervous system disorders) | 0 (0) | 1 (2) — Decreased Sense of Taste
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (6)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3)
Allergic Reaction (Immune system disorders) | 0 (0) | 4 (45)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (3) — (SOB/Tachycardia/Rigors treated in ED and hospitalized)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (6)
Back Pain (General disorders) | 0 (0) | 1 (3)
Balance Impairment (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Bleeding from inguinal lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (11)
Blood in Urine (General disorders) | 0 (0) | 1 (1)
Bloody Discharge (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (11)
Colitus (General disorders) | 0 (0) | 1 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Dry Skin on eyelids
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Elevated Creatinine (Investigations) | 0 (0) | 1 (4)
Eye Disorders (Eye disorders) | 0 (0) | 1 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (10)
Hot Flashes (Vascular disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased Urinary Frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (6)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6)
Left Groin Pain (General disorders) | 0 (0) | 1 (2)
Leukocytosis (Infections and infestations) | 0 (0) | 1 (1)
Loose Stools (Gastrointestinal disorders) | 0 (0) | 1 (4)
LUE + LLE Swelling (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms Benign, Malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Paper Cut Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Paper cut that resulted in a bullous type infection
Paresthesia (Nervous system disorders) | 0 (0) | 1 (9)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Rash (Upper Back) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5)
Rathke's Cyst (Pituitary) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Red blotches upper + lower trunk (General disorders) | 0 (0) | 1 (3)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Throat Tightness (General disorders) | 0 (0) | 1 (4)
Tremor (Nervous system disorders) | 0 (0) | 1 (3)
Trigeminal Nerve Disorder (Nervous system disorders) | 0 (0) | 1 (3)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (3)
Watery Stool (Colitis) (Gastrointestinal disorders) | 0 (0) | 1 (3)
Worsening Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)

LIMITATIONS AND CAVEATS:
Study was closed prematurely due to study supporter decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03719131/Prot_SAP_000.pdf